CLINICAL TRIAL: NCT06136364
Title: Open-label, Dose-escalation Phase 1 Clinical Study of SENL101 Autologous T Cell Injection in the Treatment of Adult Patients With Relapsed or Refractory T-LBL/ALL
Brief Title: CD7 CAR-T in Adults With Relapsed or Refractory T-LBL/ALL Clinical Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: senlangbio
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: T-lymphoblastic Lymphoma; T-ALL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD 7 CAR-T (Experimental)
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — CAR-T immunotherapy targeting CD7+

SUMMARY:
To evaluate the tolerability and safety of SENL101 in patients with relapsed or refractory T-LBL/ALL.

DETAILED DESCRIPTION:
Main research purposes:

To evaluate the tolerability and safety of SENL101 in patients with relapsed or refractory T-LBL/ALL.

Secondary research purposes:

To preliminarily evaluate the efficacy, pharmacokinetics and pharmacodynamics of SENL101 in the treatment of patients with relapsed or refractory T-LBL/ALL.

Exploratory research purpose：

1. To explore the immunogenicity of SENL101；
2. T cell NK cell recovery time after treatment；

ELIGIBILITY:
Inclusion Criteria:

According to the WHO hematopoietic and lymphoid tissue tumors classification, Subjects with refractory/relapsing T-LBL/ALL has been adequately treated and there is a lack of effective treatment, met one of the following criteria:

1. relapse: Primordial cells (>5%)in peripheral blood or bone marrow appeared again after complete remission with standard treatment or Extramedullary disease appears，include：

   1. Early recurrence within 12 months，
   2. Late recurrence at 12 months or above and with no remission after a course of standard induction chemotherapy，
   3. Recurrence after autologous or allogeneic hematopoietic stem cell transplantation ;
2. Refractory: patients who have received at least two courses standard induction regimen and failed to achieve a complete response or complete remission was not achieved after first-line or above salvage treatment;
3. The tumor cells detected by bone marrow flow cytometry were CD7+ and/or extramedullary lesions were diagnosed as CD7+ by pathological immunohistochemistry at the time of enrollment and screening;
4. If tumor cells were detected in peripheral blood during enrollment and screening, it was required to meet the requirement that the surface immunophenotype of tumor cells was CD4 and CD8 double negative by flow cytometry.
5. Life expectancy greater than 12 weeks;
6. ECOG 0-2;
7. Age 18-75 (upper and lower limits included);
8. HGB at least 70g/L,PLT 50x109/L, can be transfused;
9. Liver and kidney functions The cardiopulmonary functions meet the following requirements:

   1. Oxygen saturation under air ≥ 92%;
   2. LVEF≥50%;
   3. Total bilirubin <3×ULN;
   4. ALT/AST<3×ULN;
   5. Creatinine <1.5×ULN or creatinine clearance rate(Cockroft-Gault)>50ml/min;
10. Informed consent explained to, understood by and signed by patient/ guardian.

Exclusion Criteria:

Those who meet any of the following criteria are not eligible to join the group:

1. New York Heart Association (NYHA) classification ≥ grade III heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris or other clinically prominent heart disease within one year before signing the informed consent form, Or QTc interval >480ms at screening (QTc interval calculated by Fridericia formula);
2. If the patient has a history of hematopoietic stem cell transplantation, 6 months after the patient received allogeneic hematopoietic stem cell transplantation;
3. Those with active GvHD or those who require immunosuppressive therapy;
4. Malignancy other than T-cell acute lymphoblastic leukemia/lymphoma within 5 years prior to screening, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer after radical surgery, radical surgery ductal carcinoma in situ;
5. History of non-neoplastic central nervous system disease (Seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, neuropathy)
6. Active or uncontrollable infection requiring systemic treatment within 7 days prior to screening (except for mild urogenital infections and upper respiratory tract infections);
7. History of autoimmune disease (eg, rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease) requiring systemic immunosuppressive/systemic disease modulating medication within the past 2 years;
8. When screening, if the hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HbcAb) is positive, and the peripheral blood hepatitis B virus (HBV) DNA is higher than the detection limit, it needs to be excluded; if the hepatitis C virus (HCV) antibody is positive, the peripheral blood HCV Those with positive RNA need to be excluded; those with positive human immunodeficiency virus (HIV) antibody; those with positive cytomegalovirus (CMV) DNA test; those with positive test for Treponema pallidum specific antibody (TPPA) need to be excluded;
9. Participate in other clinical trials within 4 weeks before the informed consent is signed, or the date of the informed consent is signed and the last medication of the drug is still within 5 half-lives of the drug (whichever is longer);
10. History of severe allergy to biological products;
11. Unstable systemic disease as judged by the investigator: including but not limited to severe liver, kidney or metabolic disease requiring drug therapy;
12. Pregnant or breastfeeding women, and female subjects planning pregnancy within 2 years of cell infusion or male subjects whose partner is planning pregnancy within 2 years of cell infusion;
13. Subjects who have received CAR-T therapy or other gene-modified cell therapy prior to screening;
14. Circumstances that the investigator believes may increase the risk to the subject or interfere with the results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2038-08-14 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | 28 days after infusion
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Dr, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China